CLINICAL TRIAL: NCT07048223
Title: Effects of Expiratory Muscle Training on Posture, Balance, Trunk Control, and Respiratory Function in Children With Cerebral Palsy
Brief Title: Expiratory Muscle Training in Children With Cerebral Palsy
Acronym: CP-EMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeUni-Z.KAVRIK.001
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; expiratory muscle training; trunk control; posture; balance; respiratory rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial consists of two parallel groups and is designed to compare the effects of expiratory muscle training with those of sham expiratory muscle training in children with spastic-type cerebral palsy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Muscle Training (Experimental): In this group, expiratory muscle training will be administered using the POWERbreathe EX1 device, set at 50% of each participant's measured maximal expiratory pressure (MEP). Participants will be instructed to perform the exercises daily at home for a duration of 8 weeks. Interim assessments will be conducted every 10 days. Exercise compliance will be monitored using daily exercise tracking forms.
  Interventions: Behavioral: Expiratory Muscle Training
- Sham Expiratory Muscle Training (Sham Comparator): In the sham expiratory muscle training group, participants will perform a respiratory exercise program including breathing control, diaphragmatic breathing, and thoracic expansion exercises. In addition, sham expiratory muscle training will be administered using the POWERbreathe EX1 device set at 10% of the participant's measured maximal expiratory pressure (MEP), providing minimal resistance.
  Participants will be instructed to perform the exercises daily at home for a period of 8 weeks. Compliance will be monitored through exercise tracking forms. No progressive loading or resistance adjustments will be made during the intervention period.
  Interventions: Behavioral: Sham Expiratory Muscle Training

INTERVENTIONS:
Behavioral: Expiratory Muscle Training — In the expiratory muscle training group, participants will receive a respiratory exercise program consisting of breathing control, diaphragmatic breathing, and thoracic expansion exercises. In addition, expiratory muscle training (EMT) will be performed using the POWERbreathe EX1 device at 50% of each participant's measured maximal expiratory pressure (MEP).
  Participants will be instructed to perform 25 repetitions per session, structured as 5 cycles of 5 breaths with 1-minute rest intervals between each cycle. The training will be performed daily at home for a duration of 8 weeks. Compliance will be monitored through exercise tracking forms.
  To ensure progressive loading, MEP will be reassessed every 10 days, and the resistance of the device will be adjusted accordingly. Participants will be invited for in-person interim evaluations at these 10-day intervals to update their training parameters.
  Arms: Expiratory Muscle Training
Behavioral: Sham Expiratory Muscle Training — In the sham expiratory muscle training group, participants will perform a respiratory exercise program including breathing control, diaphragmatic breathing, and thoracic expansion exercises. In addition, sham expiratory muscle training will be administered using the POWERbreathe EX1 device set at 10% of the participant's measured maximal expiratory pressure (MEP), providing minimal resistance.
  Participants will be instructed to perform the exercises daily at home for a period of 8 weeks. Compliance will be monitored through exercise tracking forms. No progressive loading or resistance adjustments will be made during the intervention period.
  Arms: Sham Expiratory Muscle Training

SUMMARY:
This study aims to examine the effects of expiratory muscle training on posture, trunk control, balance, selective motor control, and respiratory function in children with spastic-type cerebral palsy (CP). The research focuses on evaluating an innovative rehabilitation approach that addresses common challenges observed in children with CP, such as trunk instability, reduced respiratory capacity, and postural abnormalities.

In individuals with CP, the ineffective use of respiratory muscles affects not only the respiratory system but also trunk control and overall motor performance. While most existing studies emphasize inspiratory muscle training, research on expiratory muscle training remains limited. Therefore, this study seeks to fill this gap by investigating the neuromotor effects of expiratory muscle training-an emerging component of respiratory rehabilitation-in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Age between 12 and 18 years
* Gross Motor Function Classification System (GMFCS) Level I or II
* Communication Function Classification System (CFCS) Level I, II, or III
* Spasticity graded as 0, 1, 1+, or 2 on the Modified Ashworth Scale
* No history of Botulinum Toxin-A injection or orthopedic surgery within the past 6 months

Exclusion Criteria:

* Spasticity graded as 3 or 4 on the Modified Ashworth Scale Uncontrolled seizures
* Presence of congenital cardiopulmonary disease, autism spectrum disorder, balance-impairing conditions, or significant visual/hearing impairments
* Acute respiratory tract infection

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength Assessment (MIP/MEP) | Before treatment, week 8
Peak Cough Flow | before treatment, week 8
Assessment of Posture (PostureScreen App) | before treatment, week 8
Trunk Control Assessment (ProKin Star Excursion Balance Test, Trunk Control Measurement Scale (TCMS)) | Before treatment, week 8
  Trunk control will be assessed using the Trunk Control Measurement Scale (TCMS) and the ProKin Star Excursion Balance Test. The TCMS evaluates static and dynamic trunk control in children with cerebral palsy. Scores range from 0 to 58, with higher scores indicating better trunk control. The ProKin Star Excursion Balance Test measures postural stability and trunk coordination using a computerized force platform. Assessments will be conducted before treatment and at the end of the 8th week.
Balance Assessment (PROKIN®) | before treatmant, week 8
Selective Motor Control Assessment (SCALE), (Noraxon MyoMotion) | before treatment, week 8
  Selective motor control will be assessed using the Selective Control Assessment of the Lower Extremity (SCALE). The SCALE evaluates the ability to perform isolated joint movements in the lower limbs and is scored bilaterally. Each limb can score from 0 to 10 points, with a total possible score ranging from 0 to 20. Higher scores indicate better selective voluntary motor control. Additionally, Noraxon MyoMotion will be used to collect objective kinematic data to support the SCALE assessment.

SECONDARY OUTCOMES:
Communication Function Classification System (CFCS) | before treatment
  The Communication Function Classification System (CFCS) is a five-level classification system used to describe everyday communication performance in individuals with cerebral palsy. Levels range from I (most effective communicator) to V (least effective communicator). Lower levels indicate more effective and independent communication abilities.
Gross Motor Function Classification System (GMFCS) | before treatment
  The Gross Motor Function Classification System (GMFCS) is a five-level system used to classify gross motor function in children with cerebral palsy. Levels range from I (most independent) to V (most limited). Lower levels represent better motor function and greater independence in mobility.
Muscle Tone Evaluation (Modified Ashworth Scale (MAS)) | before treatment
  Muscle tone will be assessed using the Modified Ashworth Scale (MAS), a widely used clinical tool for measuring spasticity. The scale ranges from 0 to 4, with an additional score of 1+ to indicate slight increases in muscle tone. A score of 0 indicates no increase in muscle tone, while a score of 4 indicates a rigid limb in flexion or extension. Higher scores reflect greater spasticity.
Gross Motor Function Measure (GMFM) | before treatment, week 8
  Gross motor function will be evaluated using selected sections of the Gross Motor Function Measure (GMFM-88), a standardized observational tool developed to assess changes in motor function in children with cerebral palsy. In this study, only dimensions D (Standing) and E (Walking, Running, and Jumping) will be administered. Each item is scored on a 4-point ordinal scale from 0 (does not initiate) to 3 (completes the activity). Scores will be expressed as a percentage of the maximum possible score for the selected dimensions, with higher percentages indicating better gross motor performance.
Modified Functional Reach Test (MFRT) | before treatment, week 8
  Dynamic balance will be assessed using the Modified Functional Reach Test (MFRT), which evaluates the maximum distance an individual can reach forward and laterally while maintaining a fixed base of support in a seated position. The test is performed in three directions: forward, right, and left. The distance is measured in centimeters. Higher reach distances indicate better dynamic sitting balance and trunk stability.
Prone Plank Test | before treatment, week 8
  Core endurance will be assessed using the Prone Plank Test, which measures the amount of time an individual can maintain a prone plank position (forearms and toes supporting the body, body in a straight line) without losing form. The test is performed on a flat surface, and time is recorded in seconds. A longer duration indicates greater core muscle endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek ÇOKAR, Study Chair — Istinye University

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guideline.

REFERENCES:
- [Background] de Lima Crispim TR, Neto MG, Crispim TRL, Dias RB, de Albuquerque MDM, Saquetto MB, Magalhaes PAF. Addition of respiratory exercises to conventional rehabilitation for children and adolescents with cerebral palsy: a systematic review and meta-analysis. World J Pediatr. 2023 Apr;19(4):340-355. doi: 10.1007/s12519-022-00642-1. Epub 2022 Nov 15. PMID 36376558
- [Background] Menezes KKP, Avelino PR, Alvarenga MTM, Nascimento LR. Inspiratory Training for Improving Respiratory Strength, Pulmonary Function, and Walking in Cerebral Palsy: A Meta-Analysis. Pediatr Phys Ther. 2024 Apr 1;36(2):207-215. doi: 10.1097/PEP.0000000000001092. Epub 2024 Mar 29. PMID 38568267
- [Background] Ishida H, Suehiro T, Watanabe S. Comparison of abdominal muscle activity and peak expiratory flow between forced vital capacity and fast expiration exercise. J Phys Ther Sci. 2017 Apr;29(4):563-566. doi: 10.1589/jpts.29.563. Epub 2017 Apr 20. PMID 28533585